CLINICAL TRIAL: NCT04430088
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Study to Evaluate the Efficacy and Safety of VVZ-149 Injections for the Treatment of Postoperative Pain Following Bunionectomy
Brief Title: Phase 3 Efficacy and Safety Study of VVZ-149 Injections for Postoperative Pain Following Bunionectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vivozon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VVZ149-POP-P3-US005
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VVZ-149 Injections (Experimental)
  Interventions: Drug: VVZ-149 Injections
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149 Injections — IV infusion of 1000 mg of VVZ-149
  Arms: VVZ-149 Injections
Drug: Placebo — IV infusion of 0 mg of VVZ-149
  Arms: Placebo

SUMMARY:
The purpose of this phase 3 study is to evaluate the efficacy and safety of an analgesic drug candidate, VVZ-149 Injections for treating post-operative pain following bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women must be at least 18 years of age. Female subjects must meet additional criteria in relation to childbearing potential.
* Subjects must be undergoing a planned first metatarsal bunionectomy with osteotomy and internal fixation (Austin bunionectomy) without collateral procedures.
* Subjects must have the ability to provide written informed consent.
* Subjects must have the ability to understand study procedures and communicate clearly with the Investigator and staff.

Key Exclusion Criteria:

* Subjects undergoing emergency or unplanned surgery.
* Subjects who had any previous bunionectomy procedure on either foot.
* Subjects with pre-existing conditions (other than bunion) causing preoperative pain at the site of surgery.
* Female subjects who are pregnant or breastfeeding.
* Diagnosis of chronic pain and ongoing or frequent use of pain medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Time-weighted Sum of Pain Intensity Difference (SPID) from baseline over 12 hours after the start of study drug infusion (i.e., post-dose) | 0-12 hours post-dose
  Using Numeric Pain Rating Scale (NRS, 0-10)

SECONDARY OUTCOMES:
Time to onset of perceptible pain relief using the double stopwatch method | 0-12 hours post-dose
Total number of rescue medication request between 0-12 hours post-dose | 0-12 hours post-dose
Proportion of patients with >40% improvement in pain from baseline to 6 hours post-dose | 0-6 hours post-dose
Proportion of patients who take prescription opioid after discharge | 2 weeks after discharge

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Arizona Clinical Trial Site, Phoenix, Arizona
  - California Clinical Trial Site, Anaheim, California
  - Texas Clinical Trial Site, San Antonio, Texas